CLINICAL TRIAL: NCT06886477
Title: Exploring the Mediterranean Diet as A Promising Approach for Alleviating Chronic Pain in Sickle Cell Disease
Brief Title: Sickle Cell, Pain and Mediterranean Diet
Acronym: MedSCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0041
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell; Sickle Cell Disease; Sickle Cell Disease Without Crisis; Mediterranean Diet
Keywords: sickle cell; sickle cell disease; sickle cell pain; diet; Mediterranean diet
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mediterranean Diet (Experimental): Commercially prepared foods will be provided.
  Interventions: Other: Mediterranean Diet; Other: Usual Diet
- Usual Diet (Active Comparator): Consume their typical at-home diet.
  Interventions: Other: Mediterranean Diet; Other: Usual Diet

INTERVENTIONS:
Other: Mediterranean Diet — Mediterranean Diet foods will be provided for 4 weeks.
Other: Usual Diet — Participants will consume their typical at home-diet.

SUMMARY:
The goal of this study is to compare pain levels in individuals with Sickle Cell Disease while following the Mediterranean Diet to pain levels while following their usual diet.

DETAILED DESCRIPTION:
This is an exploratory, randomized, crossover-controlled feeding study of a 4-week Mediterranean Diet or usual diet control among 24 adults with sickle cell disease and chronic pain (30 will be recruited, with an estimated 24 participants completing the study).

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease Diagnosis
* Chronic non-vaso-occlusive pain experienced on average ≥ 3 days per week for > 6 months (based on a response of "Most days," "Every day," or "Some days" and not "Never" to the question "In the past 6 months, how often have you had pain?")
* Ability to speak, read, write, and understand English
* A Mediterranean Eating Pattern for Americans (MEPA-III) score <13, indicating that they do not follow a Mediterranean diet.

Exclusion Criteria:

* Having taken systemic antimicrobials (to treat an infection in the previous 4 weeks)
* History of colon cancer or inflammatory bowel disease (given potential untoward effects on the gut microbiome)
* History of Clostridium difficile infection in the preceding 12 weeks; (4) unable to agree to maintain physical activity at the current level for the duration of the study
* Currently following a Mediterranean diet, vegan diet, or dietary restrictions (e.g., religious, food intolerance/allergy) that preclude adoption of a Mediterranean diet
* Lack of access to a space to safely store and reheat food items
* Living in a facility that provides meals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum and Fecal Short Chain Fatty Acids | Baseline and day 27 or 28 of each diet
  Mass spectrometry methods for butyrate, propionate, acetate
Serum and Fecal Bile Acid Metabolites | Baseline and day 27 or 28 of each diet
  Mass spectrometry methods for primary and secondary bile acid derivatives

SECONDARY OUTCOMES:
Gut Microbiota Composition | Baseline and day 27 or 28 of each diet
  16S rRNA amplicon
Chronic Pain | Baseline and day 27 or 28 of each diet
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Survey will be used to measure the experience of chronic pain on a 1-10 scale. The higher the number, the greater the chronic pain experience.
Diet adherence | Daily up to 4 weeks during the Mediterranean diet intervention
  Checklist- participants will keep a checklist of foods consumed during the Mediterranean diet intervention period.
Diet adherence | Daily up to 4 weeks during the Mediterranean diet intervention
  Photos of uneaten foods will be texted to researchers to see which foods were not consumed.
Diet adherence | Baseline and day 27 or 28 of each diet
  Skin carotenoid concentration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided